CLINICAL TRIAL: NCT05547152
Title: Evaluation of the Effectiveness of Virtual Reality Self-rehabilitation in the Treatment of Facial Paralysis and Synkinesis
Acronym: RéMiFaSy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PI2019_843_0100
Record Dates: First submitted 2022-09-06; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Peripheral Facial Palsy; Rehabilitation; Virtual Reality
Keywords: Peripheral Facial Palsy; rehabilitation; virtual reality
MeSH Terms: interventions — Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): patients benefiting from rehabilitation associated with virtual reality
  Interventions: Other: massages; Other: motor stimulation and stretching; Other: virtual reality
- Control arm (Active Comparator): patients benefiting from rehabilitation without virtual reality
  Interventions: Other: massages; Other: motor stimulation and stretching

INTERVENTIONS:
Other: massages — The experimental rehabilitation protocol includes massages
Other: motor stimulation and stretching — motor stimulation and stretching
Other: virtual reality — Patient watches an avatar of his face performing different movements on a screen, and will have to imagine performing these movements without actually doing them.
  Arms: Experimental arm

SUMMARY:
Peripheral facial palsy affects 15 to 40 people per 100,000 inhabitants and induces important functional and social repercussions. Synkinesis is a frequent after-effect of facial palsy recovery, consisting of involuntary facial spasms that disturb the gestural harmony and can go as far as a painful hypertonic spasm. More than 55% of patients recovering from facial palsy will develop transient or permanent synkinesis. These facial hypertonias have two main causes: imperfect axonal regeneration, which is all the more important as the damage is proximal, and hyperexcitability of the facial nerve nucleus due to a lack of central control. Management is therefore essential for the functional restoration of the face, especially since synkinesis do not evolve spontaneously. The main treatments are currently botulinum toxin injection, acting on the motor plate, and functional rehabilitation, consisting on local muscle relaxation and central motor control work. In recent years, therapies based on biofeedback and acting on central motor control have shown interesting results, and technological advances in virtual reality have made it possible to deepen this treatment in patients suffering from stroke, limb trauma or Parkinson's disease. In this project, the investigators evaluate the contribution of virtual reality to the management of facial palsy, and hypothesize that self-rehabilitation using this technology will improve motor control of the skin muscles and reduce complications related to their hypertonia such as synkinesis.

ELIGIBILITY:
Inclusion Criteria:

* Patient with recent onset peripheral facial palsy (≤ 12 months).
* Patient with peripheral facial palsy of grade ≥ III on the House & Brackmann score
* Patient of legal age (≥ 18 years)
* Patient with appropriate information and informed consent

Exclusion Criteria:

* Patient with central facial palsy
* Patient with peripheral facial palsy of > 12 months onset
* Patient with peripheral facial palsy of grade < III House & Brackmann score
* Patient who has previously undergone palliative surgery
* Patient undergoing a botulinum toxin injection protocol
* Patients benefiting from enhanced protection, i.e. minors, persons deprived of their liberty by a judicial or administrative decision, persons staying in a health or social institution, adults under legal protection, pregnant or breast-feeding women and patients in emergency situations
* Patients who have not provided informed consent
* Patients with cognitive disorders that do not allow them to follow the proposed self-education protocol
* Blind or visually impaired patients (visual acuity of the better eye after correction ≤ 4/10)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-06 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
variation of number of involuntary facial spasm between both groups of patients | 12 months
  variation of synkinesis in patients with recent onset (≤ 12 months) peripheral facial palsy compared with the conventional rehabilitation protocol

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France

IPD SHARING:
Plan to Share IPD: No